CLINICAL TRIAL: NCT02129660
Title: A Phase 2, Randomized, Double-Blind Vehicle-Controlled Comparator Study of the Effect of Glycopyrrolate and Glycopyrronium in Subjects With Axillary Hyperhidrosis
Brief Title: Comparator Study of the Effect of Glycopyrrolate and Glycopyrronium in Subjects With Axillary Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Journey Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRM04-HH02
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose 1 of glycopyrrolate, 2.0% QD (Experimental): glycopyrrolate Topical Wipes
  Interventions: Drug: Dose 1 of glycopyrrolate, 2.0% QD
- Dose 2 of glycopyrrolate, 3.0% QD (Experimental): glycopyrrolate Topical Wipes
  Interventions: Drug: Dose 2 of glycopyrrolate, 3.0% QD
- Dose 1 of glycopyrronium, 2.5% QD (Active Comparator): glycopyrronium Topical Wipes
  Interventions: Drug: Dose 1 of glycopyrronium, 2.5% QD
- Dose 2 of glycopyrronium, 3.75% QD (Active Comparator): glycopyrronium Topical Wipes
  Interventions: Drug: Dose 2 of glycopyrronium, 3.75% QD
- Vehicle (Placebo Comparator): Vehicle Topical Wipes
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: Dose 1 of glycopyrrolate, 2.0% QD — Dose 1 of glycopyrrolate Topical Wipes
  Other Names: DRM04B
  Arms: Dose 1 of glycopyrrolate, 2.0% QD
Drug: Dose 2 of glycopyrrolate, 3.0% QD — Dose 2 of glycopyrrolate Topical Wipes
  Other Names: DRM04B
  Arms: Dose 2 of glycopyrrolate, 3.0% QD
Drug: Dose 1 of glycopyrronium, 2.5% QD — Dose 1 of glycopyrronium Topical Wipes
  Other Names: DRM04
  Arms: Dose 1 of glycopyrronium, 2.5% QD
Drug: Dose 2 of glycopyrronium, 3.75% QD — Dose 2 of glycopyrronium Topical Wipes
  Other Names: DRM04
  Arms: Dose 2 of glycopyrronium, 3.75% QD
Other: Vehicle — Vehicle Topical Wipes
  Arms: Vehicle

SUMMARY:
The purpose of the study is to assess the safety of 2 doses of glycopyrrolate compared to 2 doses of glycopyrronium and vehicle (5 treatment arms) for the treatment of axillary hyperhidrosis when applied once daily for 4 weeks followed by a 2-week post-dose period.

DETAILED DESCRIPTION:
This is a randomized, double-blind, vehicle controlled, parallel group, comparator study designed to assess the safety, efficacy and pharmacokinetics of two doses of glycopyrrolate compared to two doses of glycopyrronium compared to vehicle, 5 treatment arms.

Efficacy will be assessed through gravimetric assessment of sweat production using Patient Reported Outcome and the Hyperhidrosis Disease Severity Score (HDSS).

Safety will be assessed through adverse events, local skin responses, serum chemistry and hematology laboratory testing, ECGs, physical examination and vital signs.

PK blood samples will be taken study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older.
* Primary, axillary hyperhidrosis of at least 6 months duration.
* Hyperhidrosis Disease Severity Score (HDSS) of 3 or 4 at baseline.
* For each axilla, a baseline gravimetric measurement of sweat production of at least 50 mg over 5 minutes, while at rest, at room temperature.
* Male or non-pregnant, non-lactating females.

Exclusion Criteria:

* Current pregnancy or lactation.
* Prior surgical procedure for hyperhidrosis.
* Any prior axillary treatment with an anti-hyperhidrosis medical device
* Any prior treatment with an investigational drug within 4 weeks prior to Baseline/Day 1 or within 5 elimination half lives of the active agent, whichever is longer or 6 weeks if the elimination half life is not known. Experimental devices are excluded without the approval of the Medical Monitor.
* Prior treatment with botulinum toxin (e.g., Botox®) for axillary hyperhidrosis within 1 year of Baseline/Day 1.
* Subjects with clinically significant abnormalities in laboratory values.
* Subjects with a positive Hepatitis or HIV.Hepatitis B surface antibody positive is allowed only if the subject has a history of having received Hepatitis B vaccination and there are no clinically significant abnormalities in screening liver function tests.
* Treatment with cholinergic, serotonergic antagonists, and dopamine partial agonists thought to relieve antidepressant-induced hyperhidrosis, within one month prior to Baseline/Day 1.
* Treatment with psychotherapeutic medications for less than 4 months prior to Baseline/Day 1.
* Treatment with topical or systemic anticholinergics, adrenergic agonists (clonidine), or beta-blockers within 4 weeks of the baseline visit
* Prior treatment with axillary iontophoresis within 4 weeks of Baseline/Day 1.
* Any previous IV or oral treatment with the study drug.
* Prior treatment with the topical study drug in a previous trial.
* Axillary use of nonprescription or prescription antiperspirants within 2 weeks of study enrollment.
* Presence of a condition, within 10 years of enrollment, that may cause secondary hyperhidrosis
* Menopausal women who have had symptoms of menopause such as sweating or flushing within 3 years of the study may not be enrolled.
* Known history of Sjögren's syndrome or Sicca syndrome.
* History of glaucoma, inflammatory bowel disease, toxic megacolon, or febrile illness.
* Men with a history of urinary retention requiring catheterization due to prostatic hypertrophy or severe obstructive symptoms of prostatic hypertrophy.
* Abnormal findings on screening ECG deemed clinically significant by the Investigator.
* History or presence of ventricular arrhythmias, atrial fibrillation, atrial flutter. History of other supraventricular tachycardia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne M. Deans, MT, Study Director — Dermira, Inc.
Locations (15):
- United States (14):
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Center For Dermatology Clinical Research, Fremont, California
  - Olympian Clinical Research, Tampa, Florida
  - Kenneth R. Beer MD, West Palm Beach, Florida
  - Shideler Clinical Research Center, Carmel, Indiana
  - Saint Louis University Dermatology, St Louis, Missouri
  - Haber Dermatology and Cosmetic Surgery, Beachwood, Ohio
  - Rivergate Dermatology Clinical Research Center, PLLC, Goodlettsville, Tennessee
  - DermResearch, Inc, Austin, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Dermatology Associates, Seattle, Washington
  - Women's Clinical Research Center, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington
- Innovaderm Research Inc., Montreal, Canada

REFERENCES:
- [Derived] Pariser DM, Lain EL, Mamelok RD, Drew J, Mould DR. Limited Systemic Exposure with Topical Glycopyrronium Tosylate in Primary Axillary Hyperhidrosis. Clin Pharmacokinet. 2021 May;60(5):665-676. doi: 10.1007/s40262-020-00975-y. Epub 2021 Jan 12. PMID 33433785

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose 1 of Glycopyrrolate: Dose 1 of glycopyrrolate Topical Wipes
- Dose 2 of Glycopyrrolate: Dose 2 of glycopyrrolate Topical Wipes
- Dose 1 of Glycopyrronium: Dose 1 of glycopyrronium Topical Wipes
- Dose 2 of Glycopyrronium: Dose 2 of glycopyrronium Topical Wipes
Period: Overall Study
Arm/Group | Dose 1 of Glycopyrrolate | Dose 2 of Glycopyrrolate | Dose 1 of Glycopyrronium | Dose 2 of Glycopyrronium | Vehicle
Started | 21 | 20 | 22 | 20 | 22
Completed | 19 | 20 | 21 | 20 | 20
Not Completed | 2 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose 1 of Glycopyrrolate | Dose 2 of Glycopyrrolate | Dose 1 of Glycopyrronium | Dose 2 of Glycopyrronium | Vehicle | Total
Number analyzed (Participants) | 21 | 20 | 22 | 20 | 22 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1 | 3 | 0 | 5
  Between 18 and 65 years | 21 | 19 | 21 | 16 | 22 | 99
  >=65 years | 0 | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 7 | 13 | 13 | 48
  Male | 13 | 13 | 15 | 7 | 9 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 3 | 0 | 0 | 5
  Not Hispanic or Latino | 20 | 19 | 19 | 20 | 22 | 100
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 3 | 3 | 2 | 11
  White | 18 | 20 | 16 | 17 | 20 | 91
  More than one race | 0 | 0 | 3 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Have a Minimum 2-grade Improvement in HDSS From Baseline at Week 4
Description: HDSS is a disease specific diagnostic tool that provides a qualitative measure of the severity of the subjects' condition based on how it affects daily activities.
  1 (Best), 2, 3, 4 (Worst)
Time Frame: Baseline - Week 4/ET
Population: Participant
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 of Glycopyrrolate | Dose 2 of Glycopyrrolate | Dose 1 of Glycopyrronium | Dose 2 of Glycopyrronium | Vehicle
Number analyzed (Participants) | 21 | 20 | 22 | 20 | 22
Participants | 10 | 10 | 9 | 10 | 6

2. Primary Outcome: Percentage of Subjects Who Have a Minimum 1-grade Improvement in HDSS From Baseline at Week 4
Time Frame: Baseline - Week 4
Population: Participant
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 of Glycopyrrolate | Dose 2 of Glycopyrrolate | Dose 1 of Glycopyrronium | Dose 2 of Glycopyrronium | Vehicle
Number analyzed (Participants) | 21 | 20 | 22 | 20 | 22
Participants | 16 | 17 | 15 | 14 | 12

3. Primary Outcome: Percentage of Subjects Who Have a Minimum 1-grade Improvement in HDSS From Baseline at Week 6
Time Frame: Baseline - Week 6
Population: Participant
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 of Glycopyrrolate | Dose 2 of Glycopyrrolate | Dose 1 of Glycopyrronium | Dose 2 of Glycopyrronium | Vehicle
Number analyzed (Participants) | 21 | 20 | 22 | 20 | 22
Participants | 19 | 16 | 17 | 13 | 13

4. Primary Outcome: Absolute Change in the Gravimetrically Measured Sweat Production From Baseline to Week 4
Description: Subjects are acclimated to the environment for 30 minutes. Dry gauze is weighed. The dry gauze is then applied to the subject's axilla with the arm down by the subject's side or on their lap during the 5-minute period of sweat production. The gauze with the sweat is then weighed. The difference between the Weight of the gauze with sweat and the dry gauze is the gravimetric sweat measurement in mg/5min.
Time Frame: Baseline - Week 4
Population: Participant
Measure: Mean (Standard Deviation); unit: mg/5 min
Arm/Group | Dose 1 of Glycopyrrolate | Dose 2 of Glycopyrrolate | Dose 1 of Glycopyrronium | Dose 2 of Glycopyrronium | Vehicle
Number analyzed (Participants) | 21 | 20 | 22 | 20 | 22
mg/5 min | -104.20 (73.73) | -58.27 (31.00) | -105.28 (95.83) | -72.69 (82.48) | -53.85 (70.65)

5. Primary Outcome: Absolute Change in the Gravimetrically Measured Sweat Production From Baseline to Week 6
Time Frame: Baseline - Week 6
Population: Participant
Measure: Mean (Standard Deviation); unit: mg/5 min
Arm/Group | Dose 1 of Glycopyrrolate | Dose 2 of Glycopyrrolate | Dose 1 of Glycopyrronium | Dose 2 of Glycopyrronium | Vehicle
Number analyzed (Participants) | 21 | 20 | 22 | 20 | 22
mg/5 min | -92.20 (74.87) | -44.37 (40.92) | -96.98 (103.38) | -66.17 (78.96) | -71.06 (64.82)

6. Secondary Outcome: Percentage of Subjects Who Had at Least 50% Reduction in Gravimetrically Measured Sweat Production From Baseline at Week 4
Time Frame: Baseline - Week 4
Population: Participant
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 of Glycopyrrolate | Dose 2 of Glycopyrrolate | Dose 1 of Glycopyrronium | Dose 2 of Glycopyrronium | Vehicle
Number analyzed (Participants) | 21 | 20 | 22 | 20 | 22
Participants | 19 | 16 | 20 | 16 | 15

7. Secondary Outcome: Percentage of Subjects Who Had at Least 50% Reduction in Gravimetrically Measured Sweat Production From Baseline at Week 6
Time Frame: Baseline - Week 6
Population: Participant
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 of Glycopyrrolate | Dose 2 of Glycopyrrolate | Dose 1 of Glycopyrronium | Dose 2 of Glycopyrronium | Vehicle
Number analyzed (Participants) | 21 | 20 | 22 | 20 | 22
Participants | 15 | 15 | 17 | 16 | 14

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The Total Participants at risk are based on the Safety population, defined as, Participants who were randomized and received at least one confirmed dose of study drug.
Arm/Group | Dose 1 of Glycopyrrolate | Dose 2 of Glycopyrrolate | Dose 1 of Glycopyrronium | Dose 2 of Glycopyrronium | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/22 | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/22 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 4/21 | 8/20 | 11/22 | 10/20 | 6/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose 1 of Glycopyrrolate (N=21) | Dose 2 of Glycopyrrolate (N=20) | Dose 1 of Glycopyrronium (N=22) | Dose 2 of Glycopyrronium (N=20) | Vehicle (N=21)
Mydriasis (Eye disorders) | 1 | 1 | 1 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 3 | 4 | 6 | 5 | 1
Application Site Pain (General disorders) | 0 | 1 | 0 | 1 | 5
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Accidental Exposure to Product (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Decrease Appetite (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Drug Interaction (General disorders) | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 3 | 1 | 0
Hypohidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Injection Site Bruising (General disorders) | 0 | 1 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Ocular Hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes